CLINICAL TRIAL: NCT05167552
Title: Treatment of Patients With Allergic Rhinitis and Chronic Polypous Rhinosinusitis With Olfactory Mucosa-derived Mesenchymal Stem Cells
Brief Title: Treatment of Allergic Rhinitis and Chronic Polypous Rhinosinusitis With Olfactory Mucosa-derived Mesenchymal Stem Cells
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: The Republican Center for Research and Practice in Otolaryngology (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_AllRhin
Record Dates: First submitted 2021-11-29; First posted 2021-12-22 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Allergic Rhinitis; Rhinosinusitis Chronic
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients with allergic rhinitis receiving standard treatment and mesenchymal stem cells (Experimental): Group 1: Patients with allergic rhinitis receiving standard treatment and olfactory mucosa-derived mesenchymal stem cells
  Interventions: Biological: Olfactory mucosa-derived mesenchymal stem cells; Other: Standard treatment of type Allergic Rhinitis according to the clinical protocols
- Patients with chronic rhinosinusitis receiving standard treatment and mesenchymal stem cells (Experimental): Group 2: Patients with chronic polypous rhinosinusitis receiving standard treatment and olfactory mucosa-derived mesenchymal stem cells
  Interventions: Biological: Olfactory mucosa-derived mesenchymal stem cells; Other: Standard treatment of type Chronic Polypous Rhinosinusitis according to the clinical protocols
- Patients with allergic rhinitis receiving standard treatment (Active Comparator): Group 3: Patients with allergic rhinitis receiving standard treatment
  Interventions: Other: Standard treatment of type Allergic Rhinitis according to the clinical protocols
- Patients with chronic polypous rhinosinusitis receiving standard treatment (Active Comparator): Group 4: Patients with chronic polypous rhinosinusitis receiving standard treatment
  Interventions: Other: Standard treatment of type Chronic Polypous Rhinosinusitis according to the clinical protocols

INTERVENTIONS:
Biological: Olfactory mucosa-derived mesenchymal stem cells — Olfactory mucosa-derived mesenchymal stem cells
  Arms: Patients with allergic rhinitis receiving standard treatment and mesenchymal stem cells; Patients with chronic rhinosinusitis receiving standard treatment and mesenchymal stem cells
Other: Standard treatment of type Allergic Rhinitis according to the clinical protocols — Standard treatment of type Allergic Rhinitis according to the clinical protocols
  Arms: Patients with allergic rhinitis receiving standard treatment; Patients with allergic rhinitis receiving standard treatment and mesenchymal stem cells
Other: Standard treatment of type Chronic Polypous Rhinosinusitis according to the clinical protocols — Standard treatment of type Chronic Polypous Rhinosinusitis according to the clinical protocols
  Arms: Patients with chronic polypous rhinosinusitis receiving standard treatment; Patients with chronic rhinosinusitis receiving standard treatment and mesenchymal stem cells

SUMMARY:
Treatment of patients with allergic rhinitis and chronic polypous rhinosinusitis with olfactory mucosa-derived mesenchymal stem cells

DETAILED DESCRIPTION:
During the implementation of the project, the methods for the treatment of allergic rhinitis and chronic polypous rhinosinusitis with olfactory mucosa-derived mesenchymal stem cells will be developed.

The positive outlook for the effectiveness of MSCs is due to the following:

* knowledge of the leading role of immunopathogenetic mechanisms in the development of allergic rhinitis and chronic polypous rhinosinusitis and the pronounced immunomodulating properties of MSCs;
* the ability of MSCs to reduce the production of proinflammatory cytokines and suppress immune inflammation;
* positive results of preclinical studies of the method of treatment of diseases accompanied by over-activation of the immune system, including autoimmune diseases, in animals and the first clinical studies in patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of allergic rhinitis or chronic polyposis rhinosinusitis
* The patient can read, understand, follow the examination procedures and complete, if necessary, the required documentation
* Written informed consent

Exclusion Criteria:

* The presence of any malignant tumor within the last 5 years
* Acute or chronic diseases in the stage of decompensation
* Chronic infectious diseases: HIV, viral hepatitis B, C, tuberculosis
* Patients who are pregnant, breastfeeding, or fertile patients who are not using adequate contraceptive methods
* Chronic and protracted mental disorders, all diseases with the presence of the syndrome of dependence on alcohol, drugs and psychoactive substances, any other condition that makes the patient unable to understand the nature, extent and possible consequences of the study or, in the opinion of the researcher, prevents the patient from observing and performing protocol
* Patients are unable or unwilling to give written informed consent and / or follow research procedures
* Any other medical condition that, in the opinion of the investigator, may be associated with an increased risk to the patient or may affect the outcome or evaluation of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The relapse-free period | 6 month
  The duration of the relapse-free period
The relapse-free period | 1 year
  The duration of the relapse-free period
The need for surgical intervention | 1 year
  The need for surgical intervention
The need for the use of basic drug therapy | 6 month
  The need for the use of basic drug therapy
The need for the use of basic drug therapy | 1 year
  The need for the use of basic drug therapy
Adverse effects associated with the therapy | 1 month
  Determination of adverse effects associated with the therapy
Adverse effects associated with the therapy | 1 year
  Determination of adverse effects associated with the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Antonevich, Dr, Study Director — the Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus; Yulia Eremenko, Prof, Study Director — The Republican Center for Research and Practice in Otolaryngology

IPD SHARING:
Plan to Share IPD: No